CLINICAL TRIAL: NCT01590966
Title: Scintigraphic Detection of the Biodistribution of Tumor Necrosis Factor With a Radiolabeled Anti-TNFα in Patients With Active Rheumatoid Arthritis and Active Axial and Peripheral Spondyloarthritis
Acronym: SCINTRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/279; 2009-017998-37 (EudraCT Number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2014-12

CONDITIONS: Axial and Peripheral Spondyloarthritis; Rheumatoid Arthritis
Keywords: spondyloarthritis; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis | interventions — Radioimmunodetection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with an active inflammatory joint disease (Experimental): In total there will be 20 patients included: 5 patients with active rheumatoid arthritis, 5 patients with active early axial spondyloarthritis, 5 patients with active early peripheral spondyloarthritis and 5 patients with active ankylosing spondylitis.
  Interventions: Drug: administration of Cimzia®; Drug: Immunoscintigraphy with radiolabeled Cimzia®.

INTERVENTIONS:
Drug: administration of Cimzia® — Patients will be treated with prefilled syringes containing each 200 mg/ml Cimzia® every 2 weeks which will be administered subcutaneously (The first 3 injections, a dosage of 400mg Cimzia® subcutaneously will be administered).
Drug: Immunoscintigraphy with radiolabeled Cimzia®. — All 20 patients will undergo an immunoscintigraphy with radiolabeled Cimzia®. Certolizumab pegol (Cimzia®) is an engineered humanized monoclonal antibody Fab' fragment with specificity for human TNF-α, manufactured in E. coli. The antibody fragment is subsequently purified and conjugated with high molecular weight polyethylene glycol (PEG) (40kDa). Lyophilized Cimzia® will be conjugated with S-HYNIC (a bifunctional chelator). The conjugate will be radiolabeled with Tc-99m by adding 0.1 mg Tricine, 0.01 mg SnSO4 and 750 MBq Tc-99m pertechnetate. A dose of 750 MBq Tc-99m Cimzia® will be injected intravenously.

SUMMARY:
In this open-label monocentric explorative pilot trial the objective is to show the biodistribution of TNFα by administration of radiolabeled anti-TNFα in patients with active rheumatoid arthritis and spondylarthropathy. The anti-TNFα used in this trial is certolizumab pegol (Cimzia®), a pegylated Fab'-fragment of a monoclonal antibody with high specificity for TNFα. Certolizumab pegol will be radiolabeled with 99mTechnetium. The aim of this study is to show the TNFα triggered inflammation process in the inflamed joints, especially in patients who have very early joint damage where currently other imaging methods such as X-rays are not sensitive enough for detection.

ELIGIBILITY:
INCLUSION CRITERIA FOR RHEUMATOID ARTHRITIS PATIENTS (5 PATIENTS)

* Age between 18 and 70 years-old with documented diagnosis (clinical evaluation, x-ray hands and feet minimum 2 months before inclusion) of rheumatoid arthritis minimum 3 months and maximum 15 years according to ACR criteria 1987. At least 8 tender and 8 swollen joints with inadequate response to at least 2 disease-modifying antirheumatic drugs (DMARDs) of which one is Methotrexate (MTX). Methotrexate must have been administered at least 3 months before baseline and doses and route must be stable for at least 2 months before baseline. Minimum dosage of MTX is 10 mg weekly and maximum dosage is 25 mg weekly. HAQ (Health assessment Score) score at least 25 at baseline and DAS 28(Disease Activity Score) > 3.7 at baseline.
* All patients are biological naïve patients.
* Negative for Tuberculosis (TB) (also in history) and negative screening for TB (Mantoux test / x-ray thorax)
* Female patients must be post-menopausal for at least 1 year or must underwent surgery so that they cannot become pregnant. Women of child bearing potential must use adequate contraception throughout the study and 12 weeks after the last dose of certolizumab pegol.
* Patient need to understand the study and sign an informed consent form approved by the ethics committee before participation in this study.

INCLUSION CRITERIA FOR PATIENTS WITH AXIAL SPONDYLARTHROPATY (15 PATIENTS)

* Age between 18 and 70-years old with presence of a documented diagnosis of spondylarthropathy according to current ASAS criteria valid for all of the 3 sub-groups (early axial, early peripheral and established axial)
* 10 patients with axial SpA must fulfill current ASAS criteria for AxSpA and 5 of them need to fulfill the current modified New York criteria:

  * Chronic low back pain > 3 months and onset of age < 45 years
  * Active inflammatory injury on sacro-iliac joints on MRI. Active inflammatory injuries are defined as oedema of bone in or around the sacro-iliac joints, compatible with active injuries seen on axial SpA with STIR (short tau inversion recovery) MRI
  * Inadequate response on previously, optimal use of min 2 Non-Steroidal Anti-Inflammatory Drugs (NSAIDS) in a anti-inflammatory dosage during 3 months or a medical contra-indication for use of NSAIDs
  * BASDAI score ≥ 4
* 5 patients with peripheral SpA must have presence of clinical peripheral arthritis or enthesitis or dactylitis with active disease activity, even under a stable dose of sulfasalazine during 3 months AND presence of one of the following:

  * Psoriasis of skin
  * Inflammatory bowel disease
  * Positive HLA B27
  * sacro-iliitis on image (X-ray or MRI of the sacro-iliac joints)
* all patients are anti-TNF naive
* No active tuberculosis (in medical history as current) and negative screening for latent TB (Mantoux test and X-ray thorax).
* Female patients must be post-menopausal for at least 1 year or must underwent surgery so that they cannot become pregnant. Women of child bearing potential must use adequate contraception throughout the study and 12 weeks after the last dose of certolizumab pegol.
* Patient need to understand the study and sign an informed consent form approved by the ethics committee before participation in this study.

EXCLUSION CRITERIA FOR RHEUMATOID ARTHRITIS AND SPONDYLOARTHROPATHY PATIENTS

* Patients cannot have treatment with experimental biological and non-biological therapy in the last 3 months or 5-times the half-live prior to baseline visit
* Patients who had previously treatment with anti-TNF
* Patients who had previously treatment with rituximab and/or abatacept
* Known hypersensitivity to certolizumab pegol (Cimzia®) or one of it compounds
* Current or recent medical history of progressive uncontrolled renal, hepatic, hematological, gastro-intestinal, endocrine, pulmonary, cardial, neurological or cerebral diseases.
* Severe or life threatening infections in the last 6 months; signs of current or recent infection
* Active or latent tuberculosis: in case one or more of the 3 criteria are positive: medical history of TB, recent (< 6 months) X-ray chest or recent positive PPD skin
* Known history or current viral hepatitis B of hepatitis C
* Known HIV infection
* Malignancy or history of a malignancy
* History of lymph-proliferative disease or signs/symptoms suggestive fort his disease.
* Moderate to severe hart failure (NYHA-class III/IV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Biodistribution of Cimzia® after administration of radiolabeled Cimzia®. | at baseline
  After performing the immunoscintigraphy there will be evaluation of the correlation between visualised joint inflammation on the one hand seen by clinical examination , on MRI and on ultrasound and on the other hand seen on the immunoscintigraphy.
Percentage of remission in patients, treated with Cimzia® after 14 weeks. | After 14 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Percentage of remission in patients, treated with Cimzia® after 26 weeks. | After 26 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Percentage of remission in patients, treated with Cimzia® after 38 weeks. | After 38 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Percentage of remission in patients, treated with Cimzia® after 50 weeks. | After 50 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Duration of remission in patients, treated with Cimzia® after 14 weeks. | After 14 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Duration of remission in patients, treated with Cimzia® after 26 weeks. | After 26 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Duration of remission in patients, treated with Cimzia® after 38 weeks. | After 38 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.
Duration of remission in patients, treated with Cimzia® after 50 weeks. | After 50 weeks of administration.
  All patients will be treated with Cimzia®. A specific therapy strategy will be applied: the 10 patients with early spondyloarthropathy (axial and peripheral) that are in a clinical remission on 2 consecutive visites (= week 14, 26, 38 and 50) will stop treatment after a minimum of 26 weeks treatment. If these patients are not in a clinical remission at week 26, then they will be treated further with continuous administration. The 5 patients with active rheumatoid arthritis and 5 patients with already existing longer axial spondyloarthropathy get continuous administration.

SECONDARY OUTCOMES:
Improvement in the tender and swollen joint count. | 26 weeks after baseline.
  A secondary endpoint will be the changes in the tender and swollen joint count (76/78 joint count) at week 26 in comparison with baseline.
Improvement in enthesitis | 26 weeks after baseline.
  This will be done by using the different scoring systems with inclusion of all relevant entheses.
Improvement in global measurements of disease activity. | 26 weeks after baseline.
  patient global assessment of disease activity, patient pain assessment (peripheral and axial pain), physician global assessment of disease activity, BASDAI and DAS28.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Van den Bosch, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Carron P, Lambert B, Van Praet L, De Vos F, Varkas G, Jans L, Elewaut D, Van den Bosch F. Scintigraphic detection of TNF-driven inflammation by radiolabelled certolizumab pegol in patients with rheumatoid arthritis and spondyloarthritis. RMD Open. 2016 Jun 24;2(1):e000265. doi: 10.1136/rmdopen-2016-000265. eCollection 2016. PMID 27403334
- See also: Related Info — http://www.uzgent.be